CLINICAL TRIAL: NCT07187973
Title: A Phase 1b Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DISC-3405 in Participants With Sickle Cell Disease
Brief Title: A Phase 1b, Open-Label Study of DISC-3405 in Participants With Sickle Cell Disease (SCD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DISC-3405-102
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Up to 2 cohorts of participants are planned:
  * Cohort A will enroll 12 participants with HbSC or HbSS. At least one-third of participants must be HbSC, and at least one-third of participants must be HbSS.
  * Cohort B is optional and will enroll up to 12 participants with HbSC or HbSS, administering previously studied or lesser dose levels and regimens
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Within-participant dose escalation (Experimental): This is an open-label, multicenter, within-participant dose-escalation study examining up to 3 dose levels of DISC-3405.
  Interventions: Drug: DISC-3405

INTERVENTIONS:
Drug: DISC-3405 — DISC-3405 is administered subcutaneously.

SUMMARY:
This is an open-label, multicenter, within-participant dose-escalation study examining up to 3 dose levels of DISC-3405 and will assess the safety, tolerability, PK, and PD of DISC 3405 in participants with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at the time of signing the informed consent form (ICF).
2. Male or female study participants with SCD HbSC or HbSS.
3. Participants who have been diagnosed with any of the following SCD-related complications: between 1-10 episodes of VOC in the past 12 months, any history of sickle cell related retinopathy, silent cerebral infarct, avascular necrosis, sensorineural hearing loss; or at least 1 episode of priapism, hepatic sequestration, splenic sequestration, or splenic infarct within the last 12 months as assessed locally.
4. Hgb ≥7.0 g/dL during Screening. The first 2 participants must have an Hgb ≥9 g/dL.
5. Normal alpha globin gene screen.
6. Absolute reticulocyte count or % reticulocyte count >1.5 × upper limit of normal (ULN) during Screening.
7. TSAT ≥15% at Screening.
8. Ferritin ≥50 ng/mL for HbSC or ≥100 ng/mL for HbSS (ferritin must be <1000 ng/mL at Screening).
9. For participants taking hydroxyurea, L-glutamine, or crizanlizumab, stable dose for at least 2 months prior to Screening and with no anticipated need for dose adjustments during the study.
10. If male, not vasectomized for at least 6 months, with female sexual partner(s) of childbearing potential, agrees he and partner will use double methods of the following highly effective methods of birth control (described below) from the first dose of randomized study drug until 120 days after the last administration of study drug and must not donate sperm during their study participation:

    1. Stable hormonal contraceptive (≥3 months; female partner) in conjunction with a barrier method (eg, condom [male or female] or diaphragm).
    2. Intrauterine device, in place for at least 3 months (female partner) in conjunction with a barrier method (eg, condom [male or female] or diaphragm).
    3. Surgically sterile by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation (female partner) in conjunction with a barrier method (eg, condom [male or female] or diaphragm).
11. If female, then EITHER postmenopausal, defined as at least 12 months natural, spontaneous amenorrhea, 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) >40 mIU/mL at Screening, or at least 6 weeks following surgical menopause (bilateral oophorectomy with or without hysterectomy); surgically sterile, OR agree to use 1 of the following highly effective methods of birth control on Day 1 (or earlier) and for at least 120 days after the last administration of study drug:

    1. Stable hormonal contraceptive (≥3 months) in conjunction with a barrier method (eg, condom [male or female] or diaphragm).
    2. Intrauterine device, in place for at least 3 months in conjunction with a barrier method (eg, condom [male or female] or diaphragm).
    3. Tubal ligation or single male partner with vasectomy in conjunction with a barrier method (eg, condom [male or female] or diaphragm).
12. Negative pregnancy test (females of childbearing potential) prior to dosing.
13. Able to understand the study aims, procedures, and requirements, and provide written informed consent.
14. Able to comply with all study procedures.

Exclusion Criteria:

1. Participants who are receiving regularly scheduled blood (RBC) transfusion therapy or phlebotomy or have received RBC transfusion or phlebotomy within 60 days of Screening.
2. Hospitalized for VOC or other sickle cell related complication within 14 days of Screening.
3. Participants with clinically significant bacterial, fungal, parasitic, or viral infection.
4. Active HIV, hepatitis B, or C. A positive hepatitis or HIV result should be discussed between the Investigator and Sponsor prior to enrollment.
5. Significant renal dysfunction, evidenced by estimated glomerular filtration rate of <60 mL/min/1.73 m2 at the Screening visit, as assessed locally.
6. Hepatic dysfunction characterized by alanine aminotransferase (ALT) >2.5 × ULN.
7. Any episode of ACS in the last 6 months.
8. Prior or planned hematopoietic stem cell transplant or gene therapy.
9. History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to Screening.
10. History of invasive malignancies within the last 5 years, except localized cured prostate cancer and cervical cancer, or other malignancies deemed acceptable by the Sponsor.
11. Major surgery within 8 weeks before Screening or incomplete recovery from any previous surgery.
12. A history or known allergic reaction to any IP excipients or history of anaphylaxis to any food or drug.
13. History of alcohol dependence or excessive alcohol consumption, as assessed by the Investigator.
14. Other medical or psychiatric condition or laboratory finding not specifically noted above that, in the judgment of the Investigator or Sponsor, would put the participant at an unacceptable risk or otherwise preclude the participant from participating in the study.
15. Condition or concomitant medication that would confound the ability to interpret clinical, clinical laboratory, including a major psychiatric condition that has had an exacerbation or required hospitalization in the last 6 months.
16. If female, pregnant or breastfeeding.
17. Participation in any other clinical protocol or investigational study that involves administration of experimental therapy and/or therapeutic devices within 30 days of Screening.
18. Participants with a history of transient ischemic attack or stroke may be considered in consultation with Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of DISC-3405 administration in participants with SCD | Up to 36 weeks
  Proportion of participants with treatment-emergent adverse events (TEAEs), changes in vital signs, changes in physical examinations, changes in electrocardiograms (ECGs), and changes in clinical laboratory results

SECONDARY OUTCOMES:
Pharmacodynamic (PD) properties of DISC-3405 in participants with SCD by change from baseline for hemoglobin (Hgb) | Up to 36 weeks
Pharmacodynamic (PD) properties of DISC-3405 in participants with SCD by change from baseline for hematocrit (HCT) | Up to 36 weeks
Pharmacodynamic (PD) properties of DISC-3405 in participants with SCD by change from baseline for reticulocyte count | Up to 36 weeks
Pharmacodynamic (PD) properties of DISC-3405 in participants with SCD by change from baseline for Red Blood Cell Count (RBC) | Up to 36 weeks
Pharmacodynamic (PD) properties of DISC-3405 in participants with SCD by change from baseline for Lactate Dehydrogenase (LDH) | Up to 36 weeks
Pharmacodynamic (PD) properties of DISC-3405 in participants with SCD by change from baseline for bilirubin (direct and indirect) | Up to 36 weeks
Area under the plasma concentration versus time curve (AUCt,) following the first dose | Up to 36 weeks
Area under the plasma concentration versus time curve extrapolated to infinity (AUC∞) following the first dose | Up to 36 weeks
Maximum plasma concentration (Cmax) following the first dose | Up to 36 weeks
Time to maximum plasma concentration after drug administration (Tmax) | Up to 36 weeks
Elimination half-life (T1/2el) following the first dose | Up to 36 weeks
Apparent clearance (CL/F) following the first dose | Up to 36 weeks
Pre-dose trough concentration (Ctrough) after repeating doses | Up to 36 weeks
Apparent volume of distribution corrected for bioavailability (Vd/F) | Up to 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Julie Kanter, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No